CLINICAL TRIAL: NCT06720727
Title: Craniospinal Irradiation in Histone AlteRed Midline Glioma (CHARM) - A Phase II Open Label Prospective Study
Brief Title: Craniospinal Irradiation in Histone AlteRed Midline Glioma
Acronym: CHARM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4481
Record Dates: First submitted 2024-10-30; First posted 2024-12-06 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — Craniospinal Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Craniospinal irradiation involves delivery of radiation therapy to the whole brain, spinal cord, nerve roots, the covering meninges(leptomeninges) and subarachnoid space and provides a viable means of mitigating leptomeningeal spread and possibly improving survival.
  Interventions: Radiation: craniospinal irradiation

INTERVENTIONS:
Radiation: craniospinal irradiation — Delivering radiotherapy to brain, spinal cord and its covering membrane.

SUMMARY:
Paediatric H3K27/H3G34 mutant diffuse midline gliomas are high grade gliomas that arise in midline structures/cerebral hemispheres and are known to have dismal outcomes. Standard treatment includes definitive radiation therapy to primary site along with concurrent temozolomide chemotherapy following histological confirmation with a biopsy. Studies have shown poorer outcomes in the paediatric age group compared to that of adults and an increased risk to fail/recur in the leptomeninges(covering of brain and spinal cord). The following study is planned in order to assess the benefit of craniospinal irradiation(delivering radiotherapy to brain, spinal cord and its covering membrane in this high risk population. Thereby the investigator aim to improve survival in newly diagnosed histone mutant pediatric midline gliomas in the upfront setting. Patterns of disease failure, treatment related toxicities and quality of life will also be assessed as a part of this study. If proven beneficial, this study will influence how patients with this diagnosis will be treated in the future.

DETAILED DESCRIPTION:
Introduction: Paediatric H3K27/H3G34 mutant diffuse midline gliomas (DMGs) are aggressive high-grade gliomas predominantly affecting midline structures and cerebral hemispheres. Despite aggressive therapy including radiation and chemotherapy, these tumors carry a poor prognosis, particularly in children, with frequent recurrence and high risk of leptomeningeal spread. Current standard treatment involves definitive radiation therapy to the primary site and concurrent temozolomide chemotherapy following histological confirmation via biopsy. However, outcomes remain suboptimal, prompting exploration of more intensive therapeutic strategies.

Primary objective:

To study if the addition of craniospinal irradiation to standard practice improves outcomes in pediatric diffuse midline glioma.

Secondary objectives:

* Estimate median time to leptomeningeal dissemination and compare with historical control
* Study patterns of failure
* Early and late toxicities
* Study quality of life indices
* To estimate QTWiST (Quality of life without symptoms or toxicity)

Primary endpoint: Overall survival at 12 months

Secondary endpoints:

* Time to leptomeningeal dissemination in months
* Incidence of different failure patterns from clinico-radiological assessment
* Toxicity assessment with the NCI Common Terminology Criteria for Adverse Events version 5 (CTCAE v5) during CSI(weekly), at conclusion of radiotherapy , post completion of 6 cycles adjuvant temozolomide, and in subsequent follow-ups at 3, 6, 9 and 12 months.
* Quality of life indices using the EORTC QLQC- 30 and its BN -20 module at baseline, after completion of radiotherapy, post completion of 6 cycles adjuvant temozolomide and in subsequent follow-up visits at 3, 6, 9 and 12 months.
* Quality of life without symptoms or toxicity in three health states TOX (toxicity), TWIST (time without symptoms) and REL (relapse) at baseline, after completion of radiotherapy, post completion of 6 cycles adjuvant temozolomide and in subsequent follow-up visits at 3, 6, 9 and 12 months.

Study setting: The study will be conducted in the department of Radiation Oncology, Neuro Oncology Disease management group

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed biopsy proven histone altered diffuse midline glioma
2. Age- ≥3 to <18 years at time of diagnosis
3. Karnofsky/Lansky Performance Score more than or equal to 70
4. Has provided written informed consent/ assent form
5. No prior therapy except debulking surgery or biopsy

Exclusion Criteria:

1. Recurrent or progressive disease
2. Clinical features or family history suggestive of Inherited Cancer Predisposition such as Constitutional Mismatch Repair Deficiency (CMMRD)
3. Previous history of malignancy
4. Not willing /unlikely to comply with proposed therapy and follow up

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2028-11-08 (Estimated); Study Completion 2028-11-08 (Estimated)

PRIMARY OUTCOMES:
Survival Outcomes | at 12 months
  Overall survival- time in months between the date of diagnosis to date of death due to any cause

SECONDARY OUTCOMES:
Leptomeningeal Dissemination | at 12 months
  Time to leptomeningeal dissemination (will be defined as time in months between completion of planned therapy to the date of confirmation of leptomeningeal metastasis)
Patterns of failure | at 12 months
  Incidence of different patterns of failure from diagnosis ( the time point of measurement of the primary outcome - overall survival
Any treatment emergent acute toxicity recording | Baseline , week 1 , week 2 , week 3 , week 4 , week 5 ,week 6 , conclusion of RT
  All treatment emergent acute toxicity- expected (nausea, vomiting, hematological, dermatitis and mucositis) and unexpected, will be recorded.
  Grading will be done for all using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5
Quality of life indices | will be done at 3 months
  Objective scoring with European Organisation For Research And Treatment Of Cancer(EORTC) Quality of Life Questionnaire(QLQC-30), brain specific module (BN 20)
QTWiST (Quality of life Without Symptoms or Toxicity) calculation | will be done at 3 months
  Objective score calculation using mean duration in each health state weighed by a utility coefficient; from QLQC 30- BN 20 scores and the time spent in serious toxicity and without relapse.
Any treatment emergent late toxicity recording | After completion of 6 cycles of adjuvant chemotherapy, at 3months, 6months, 9months and 12months follow up
  All treatment emergent late toxicity- expected and unexpected, will be recorded after completion of chemotherapy. Grading will be done for all using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Chatterjee, MD, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, India

IPD SHARING:
Plan to Share IPD: No